CLINICAL TRIAL: NCT04639843
Title: A Phase 1 Study of Doxorubicin, CC-486 (5-azacitidine), Romidepsin, and Duvelisib (hARD) for T-cell Lymphoma
Brief Title: Doxorubicin, CC-(486) (5-azacitidine), Romidepsin, and Duvelisib (hARD) for T-cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety issues with PI3 kinase inhibitors
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200169; 20-C-0169
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Adult T-cell Leukemia/Lymphoma; Extranodal NK-/T-cell Lymphoma, Nasal Type; Enteropathy-Associated T-Cell Lymphoma; Monomorphic Epiteliotrophic Intestinal T-cell Lymphoma; Hepatosplenic T-cell Lymphoma
Keywords: TCL; Histone Deacetylase Inhibitors (HDACi); Kinase Inhibitors
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Enteropathy-Associated T-Cell Lymphoma | interventions — cc-486; duvelisib; romidepsin; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1- Experimental Treatment: Dose Escalation (Experimental): Duvelisib (PO BID) at escalating doses of 25, 50 and 75 mg/BID on days -14 to 14 of C1 and days 1-14 of all other cycles of each 21- day cycle (max 8 cycles) with CC-486 (5-azacitidine) (PO) at 300mg/day on days 1-10, romidepsin at 12mg/m2 (IV) on Days 1 and 8 of each cycle and doxorubicin (IV) at 25 mg/ m2 on Day 1 of cycles 3-8 (Cycles 3-6 for patients with prior anthracycline-based therapy), to determine RP2D of duvelisib and doxorubicin
  Interventions: Drug: CC-486 (5-azacitidine); Drug: Duvelisib; Drug: Romidepsin; Drug: Doxorubicin
- 2 - Experimental Treatment: Dose Expansion (Experimental): Duvelisib (PO BID) at RP2D on days -14 to 14 of C1 and days 1-14 of all other 21-day cycle (max 8 cycles) with CC-486 (5-azacitidine) at 300mg/day (PO) on days 1-10, romidepsin at 12mg/m2 (IV) on days 1 and 8 of each cycle, and doxorubicin at 25 mg/m2 on day 1 of Cycles 3-8 (Cycles 3-6 for patients with prior anthracycline-based therapy
  Interventions: Drug: CC-486 (5-azacitidine); Drug: Duvelisib; Drug: Romidepsin; Drug: Doxorubicin

INTERVENTIONS:
Drug: CC-486 (5-azacitidine) — CC-486 (5-azacitidine) with a dose of 300mg oral intake daily will be given on day 1 to day 10 for 8 cycles.
Drug: Duvelisib — Duvelisib by oral intake at escalating doses of 25, 50 and 75 mg/BID on days -14 to 14 of the 1st cycle then days 1-14 of Cycles 2-8 of each 21- day cycle (max 8 cycles).
Drug: Romidepsin — Romidepsin (12mg/m2) will be administered on days 1 and 8 of each cycle through a peripheral or central intravenous catheter for 8 cycles.
Drug: Doxorubicin — Doxorubicin at 25 mg/ m2 by IV infusion on Day 1 of cycles 3-8.

SUMMARY:
Background:

T-cell lymphomas (TCLs) are rare cancers. Many types of TCLs do not develop in the lymph nodes but in places like the skin, spleen, and bone marrow. Researchers want to see if a mix of 4 drugs can help people with TCL.

Objective:

To test if the combination of romidepsin, CC-486 (5-azacitidine), duvelisib, and doxorubicin can be used safely in people with TCL.

Eligibility:

Adults 18 and older with TCL that is newly diagnosed or that returned after or did not respond to standard treatments.

Design:

Participants will be screened on a separate protocol. They may have a tumor biopsy.

Participants will have medical histories, medicine reviews, and physical exams. Their ability to do daily activities will be assessed. They will have blood and urine tests.

Participants will take duvelisib and CC-486 (5-azacitidine) by mouth. They will get romidepsin and doxorubicin by intravenous infusion. They will take the drugs for up to eight 21-day cycles. They will keep a medicine diary.

Participants will have a bone marrow aspiration and/or biopsy. Bone marrow will be taken through a needle inserted in the hip.

Participants will have tumor imaging scans. Some may have a brain MRI and lumbar puncture. Some may have skin assessments.

Participants will give blood, saliva, and tumor samples for research.

Participants will have a safety visit 30 days after treatment ends. Then they will have follow-up visits every 60 days for 6 months, then every 90 days for 2 years, and then every 6 months for 2 years. Then they will have yearly visits until their disease gets worse or they start a new treatment....

DETAILED DESCRIPTION:
Background:

T-cell lymphomas (TCLs) are a heterogeneous group of lymphoid malignancies defined by clonal proliferation of post-thymic T lymphocytes.

Patients with newly diagnosed TCLs are most commonly treated with a CHOP (cyclophosphamide, doxorubicin, vincristine and prednisone)-like regimen, with less than 30% having durable complete responses (CRs). Of the chemotherapy agents used, doxorubicin is the one which was consistently associated with prolonged progression-free survival (PFS) and overall survival (OS) in retrospective studies.

Treatment options for the 70% of patients with TCL who relapse are limited and of minimal efficacy; novel treatment strategies are urgently needed.

Many TCL have mutations in epigenetic modifier genes, and histone deacetylase inhibitors such as romidepsin are approved for treatment of peripheral T-cell lymphoma (PTCL); however, the overall response rate (ORR) with single-agent treatment is only 20-30%, and improvement in OS was not shown.

Romidepsin and the hypomethylating agent CC-486 (5-azacitidine) acted synergistically in vitro, and showed high clinical activity, with an ORR of up to 79% in some types of TCL.

Many TCLs rely on the PI3K pathway, whether through activation of CD28 through fusions or gain-of-function mutations or by interruptions of the CD28-inhibiting PD-1/PD-L1 immune checkpoint.

Duvelisib is an inhibitor of the PI3K gamma and delta isoforms; in phase I trials it has shown both single-agent activity and synergy with romidepsin for patients with TCL.

As combinations of both CC-486 (5-azacitidine)/romidepsin and duvelisib/romidepsin have demonstrated both adequate safety and clinical efficacy, safety and efficacy of the triplet combination should be explored.

Objectives:

To determine the safety and toxicity profile, maximum tolerated dose (MTD), and the recommended phase II dose (RP2D) of the four-drug combination of CC-486 (5-azacitidine), romidepsin and duvelisib, and doxorubicin, in patients with TCL.

Eligibility:

Patients with histologically or cytologically confirmed newly diagnosed or relapsed/refractory T-cell lymphoma (TCL) defined as follows:

Cohort 2: Untreated patients with any peripheral TCL, not including anaplastic large cell lymphoma (ALCL), but including acute and lymphoma subtypes of adult T-cell leukemia/lymphoma (ATLL).

Cohorts 1 and 3: Any relapsed/refractory peripheral T-cell lymphoma including ATLL and ALCL who have disease after receiving at least one line of systemic therapy, which must include brentuximab vedotin if the disease is ALCL.

Age >= 18 years of age

ECOG performance status of <= 2

Adequate organ and marrow function

Design:

Open-label, single-center, non-randomized Phase 1 study

"3 + 3" design will be used to determine the RP2D of dose-escalated duvelisib with fixed dose romidepsin CC-486 (5-azacitidine) and doxorubicin with two expansion cohorts at the RP2D

Maximum 8 cycles (21-day cycles) of combination therapy

To explore all dose levels, including further evaluation in two dose expansion cohorts, the accrual ceiling will be set at 60 patients

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients with newly diagnosed (Cohort 2) or relapsed/refractory (Cohorts 1 and 3) T-cell lymphoma (TCL) defined as follows (per 2016 WHO classification):

   * Adult T-cell leukemia/lymphoma
   * Extranodal NK-/T-cell lymphoma, nasal type
   * Enteropathy-associated T-cell lymphoma
   * Monomorphic epiteliotrophic intestinal T-cell lymphoma
   * Hepatosplenic T-cell lymphoma
   * Subcutaneous panniculitis-like T-cell lymphoma
   * Peripheral T-cell lymphoma, NOS
   * Angioimmunoblastic T-cell lymphoma
   * Follicular T-cell lymphoma
   * Nodal peripheral T-cell lymphoma with TFH phenotype
   * Anaplastic large-cell lymphoma, ALK+ and ALK- (only if relapsed/refractory after at least one line of systemic therapy, which must include brentuximab vedotin)
   * Breast implant-associated anaplastic large-cell lymphoma Note: For relapsed patients, prior treatment may include allogeneic stem cell transplantation
2. PTCL from initial diagnosis or recurrence must be histologically or cytologically proven and diagnosis be confirmed by the Laboratory of Pathology, NCI.
3. For patients without circulating lymphoma cells detectable by flow cytometry, a formalin fixed tissue block or 15 slides of tumor sample (archival or fresh) must be available at enrollment for performance of correlative studies. NOTE: Patients without circulating malignant cells must be willing to have a tumor biopsy if prior tissue or adequate archival tissue is not available (i.e., post-enrollment and prior to treatment).
4. Disease must be measurable with at least one measurable lesion by RECIL 2017 criteria or with an abnormal clonal T-cell population detectable by peripheral blood flow cytometry.
5. Age >=18 years
6. ECOG performance status <=2.
7. LVEF within institutional parameters as determined by echocardiography.
8. DLCO/VA Adjusted and FEV1 >=50% of reference.
9. Adequate organ and marrow function as defined below:

   Absolute neutrophil count >= 1,000/mcL

   Platelets >= 75,000/mcL

   Hemoglobin >= 9 g/dL (regardless of transfusion status)

   Total bilirubin <= 1.5 X institutional upper limit of normal (ULN)

   AST(SGOT)/ALT(SGPT) <= 2.5 X institutional ULN

   Creatinine clearance >= 60 mL/min/1.73 m^2 calculated by calculated using eGRF in the clinical lab
10. For women of childbearing potential (WCBP): negative serum <= human chorionic gonadotropin ( <=hCG) pregnancy test during screening. A negative pregnancy test is also required within 7 days before first treatment; screening results may be used for treatment if they fall within the required window.

    NOTE: WCBP is defined as sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months for women >55 years of age)
11. Male and female participants of reproductive potential (i.e., not surgically sterile or female subjects who are not postmenopausal), must be willing to use a highly effective method of contraception for the duration of the study treatment and 3 months after the last dose of duvelisib and/or romidepsin and for 6 months after the last dose of doxorubicin, whichever is longer.
12. For patients that have received allogeneic HSCT, a minimum of 100 days must have elapsed before enrollment. Patients must have been off of immunosuppressive medications for prophylaxis of GVHD for at least four weeks before enrollment.
13. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients who are receiving any other investigational agents.
2. Patients in need of immediate cytoreduction.
3. Chemotherapy or monoclonal antibody therapy within 4 weeks prior to start of treatment (6 weeks for nitrosoureas or mitomycin C); small molecule or radiation therapy within 2 weeks.
4. Prior lifetime doxorubicin therapy >= 400 mg/m^2.
5. Prior radiation therapy to chest with fields involving the heart.
6. Major surgery within 4 weeks prior to start of treatment
7. History of tuberculosis treatment within the 2 years prior to start of treatment
8. Administration of a live or live attenuated vaccine within 6 weeks prior to start of treatment, or of mRNA and adenovirus-based vaccines within 2 weeks prior to start of treatment
9. Patients who have received all of the planned study drugs - i.e., duvelisib, romidepsin, and CC-486 (5-azacitidine) - at any time point during prior treatments for TCL. Patients who have received one or two of the three drugs (alone or in combination) remain eligible.
10. Patients with previous malignant disease other than the target malignancy within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ.
11. Systemic treatment for acute or chronic graft versus host disease (GVHD) within 12 weeks of the first dose of duvelisib
12. Cohort 1 (Dose Escalation) only: history of grade 3/4 GVHD
13. Patients with active acute or chronic GVHD
14. History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function. Pulmonary function testing (PFTs) will be evaluated at screening.
15. Prior history of drug-induced colitis or drug-induced pneumonitis.
16. History of chronic liver disease or veno-occlusive disease
17. History of allergic reactions or known or suspected hypersensitivity attributed to compounds of similar chemical or biologic composition to duvelisib, romidepsin or mannitol and CC-486 (5-azacitidine).
18. Ongoing treatment with systemic steroids at a dose higher than 20 mg of prednisone (or equivalent) once daily
19. Patients with uncontrolled intercurrent illness including, but not limited to, detectable CMV or EBV viral load, and ongoing or active bacterial, fungal, or viral infection requiring systemic therapy, with the following exceptions:

    * Human immunodeficiency virus (HIV)-infected patients on effective anti- retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable and on suppressive therapy, if indicated.
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
    * Subjects on antimicrobial, antifungal, or antiviral prophylaxis.
20. History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drugs and/or predispose the subject to an increased risk of gastrointestinal toxicity.
21. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification Class II), congenital long QT syndrome, or other serious cardiac arrhythmia including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min).
22. Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes.
23. Uncontrolled hypertension, i.e., blood pressure (BP) of >=160/95 at screening; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria.
24. Triplicate average baseline QTcF interval >= 480 ms during screening
25. Patients taking drugs leading to significant QT prolongation Note: A 5 half-life washout period must have elapsed following the use of these drugs prior to administration of romidepsin.
26. Concomitant use of rifampin and other strong CYP3A4 inhibitors and inducers within 2 weeks prior to start of treatment.
27. Inability to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV).
28. Other severe acute or chronic medical conditions including psychiatric conditions such as recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
29. Pregnant or lactating women. NOTE: Pregnant women are excluded from this study because based on findings in animals and its mechanism of action, duvelisib can cause fetal harm when administered to a pregnant woman. In animal reproduction studies, administration of duvelisib to pregnant rats and rabbits during organogenesis caused adverse developmental outcomes including embryo-fetal mortality. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with duvelisib, breastfeeding should be discontinued if the mother is treated with duvelisib. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 8 cycles
  Rate and severity of AEs will be summarized by grade and type of toxicity
Maximum tolerated dose (MTD) | 21 days
  Frequency (number and percentage) of treatment emergent adverse events

SECONDARY OUTCOMES:
Progression-free survival | every 2 months for 6 months, every 3 months for 2 years, every 6 months for 2 years, then annually
  The response rate will be determined and reported along with a 95% confidence interval
Overall Repsonse Rate | 8 cycles
  The response rate will be determined and reported along with a 95% confidence interval
Complete Response Rate | 8 cycles
  The response rate will be determined and reported along with a 95% confidence interval
Duration of response (DOR) | every 2 months for 6 months, every 3 months for 2 years, every 6 months for 2 years, then annually
  The response rate will be determined and reported along with a 95% confidence interval
Overall Survival (OS) | every 2 months for 6 months, every 3 months for 2 years, every 6 months for 2 years, then annually
  The response rate will be determined and reported along with a 95% confidence interval
Event Free Survival (EFS) | every 2 months for 6 months, every 3 months for 2 years, every 6 months for 2 years, then annually
  The response rate will be determined and reported along with a 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0169.html